CLINICAL TRIAL: NCT00302588
Title: The Final Diagnosis and Treatment Result of Metastatic Cervical Carcinoma of Unknown Primary
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701257
Record Dates: First submitted 2006-03-12; First posted 2006-03-14 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-12

CONDITIONS: Metastasis Cervical Lymph Nodes of Unknown Primary Carcinoma
Keywords: metastatic carcinoma; cervical lymph nodes; unknown primary; diagnosis; result
MeSH Terms: conditions — Carcinoma; Disease

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
Investigate the final diagnosis and treatment result of metastatic cervical carcinoma of unknown primary

DETAILED DESCRIPTION:
Carcinoma of unknown primary (CUP) is defined as biopsy-proven metastasis of an epithelial malignancy in the absence of an identifiable primary site after complete history and physical examination, basic laboratory studies, chest X-ray and additional directed studies indicated by positive findings during the initial work-up. It is characterized by its slow local development and its high metastatic potential.1,2 Patients with CUP represent 4-10% of all new cancer patients.3,4 The presenting sites of metastasis identified pathologically, radiographically or by physical examination were found most frequently in the lymph nodes (37.1%), followed by the liver, bone, lung, pleura/pleural space, brain, peritoneum, adrenal and skin. Of the lymph nodes of metastasis, the supraclavicular cervical area is the leading site (31.3%), followed by the mediastinum, axilla, retroperitonium, and inguina.5 The incidence of metastatic cervical CUP (MCCUP) varies between 2% and 9% of all head and neck cancers.6-8 The level of cervical metastatic involvement may give some clue as to the likely primary site. A submandibular mass (level I) would most commonly be related to a primary in the oral cavity or skin. Level II nodes, including the jugulodigastric node, may point to a primary in the oral cavity, oropharynx, or supraglottic larynx. Tumours of the nasopharynx generally spread to level II or the posterior triangle, as well as retropharyngeal nodes. Middle and lower jugular nodes (levels III and IV) are more likely related to a laryngeal or hypopharyngeal cancer. Metastatic disease restricted to the supraclavicular region is often due to an infraclavicular primary site.9 The prognosis is different according to the involved lymph node level and possible primary site. Modern cancer management relies heavily on recognition of the primary tumor; thus the absence of a primary site poses major diagnostic and therapeutic problems. The patient benefits from identification of the initial tumor site because postoperative irradiation ports may be reduced and because surveillance for recurrence may be improved.10 In order to identify the likely primary site of MCCUP and compare the prognoses of known and unknown primary groups, we report the results according to the different levels of metastatic cervical lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* cases of metastatic cervical carcinoma of unknown primary

Exclusion Criteria:

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan